CLINICAL TRIAL: NCT06212102
Title: Dydrogesterone Versus GnRH Antagonist in Poor Responders Undergoing Double Ovarian Stimulation: A Randomized Controlled Non-inferiority Trial
Brief Title: Dydrogesterone Versus GnRH Antagonist in Poor Responders Undergoing Double Ovarian Stimulation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bedaya Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Double stimulation
Record Dates: First submitted 2024-01-07; First posted 2024-01-18 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Infertility
Keywords: Infertility; IVF-ET; Poor ovarian responders; Double stimulation
MeSH Terms: conditions — Infertility | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progestin primed ovarian stimulation group (Experimental): HMG ( 300IU) was used during the follicular phase of ovarian stimulation (FPS) and during the luteal phase of ovarian stimulation (LPS). Progestin (dydrogesterone) 30 mg/day was used to prevent premature LH surge during the FPS and LPS.
  In subsequent cycle, frozen embryo transfer was done
  Interventions: Drug: Progestin primed ovarian stimulation
- GnRH antagonist group (Active Comparator): HMG ( 300IU) was used during the follicular phase of ovarian stimulation (FPS) and during the luteal phase of ovarian stimulation (LPS). Flexible GnRH antagonist protocol (Cetrorelix acetate) (0.2 mg) was used to prevent premature LH surge during the FPS and LPS.
  In subsequent cycle, frozen embryo transfer was done
  Interventions: Drug: GnRH antagonist

INTERVENTIONS:
Drug: Progestin primed ovarian stimulation — HMG ( 300IU) was used during the follicular phase of ovarian stimulation (FPS) and during the luteal phase of ovarian stimulation (LPS). Progestin (dydrogesterone) 30 mg/day was used to prevent premature LH surge during the FPS and LPS.
  Arms: Progestin primed ovarian stimulation group
Drug: GnRH antagonist — HMG ( 300IU) was used during the follicular phase of ovarian stimulation (FPS) and during the luteal phase of ovarian stimulation (LPS). Flexible GnRH antagonist protocol (Cetrorelix acetate) (0.2 mg) was used to prevent premature LH surge during the FPS and LPS.
  Arms: GnRH antagonist group

SUMMARY:
The aim of this randomized controlled trial was to compare the efficacy and cost-effectiveness of using progestin with GnRH antagonist to prevent premature LH surge in poor responders undergoing double stimulation protocol.

ELIGIBILITY:
Inclusion Criteria:

Patients belonging to Poseidon group 4

Exclusion Criteria:

* PCOS
* Endometriosis
* History of recurrent abortion

Ages: 35 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Medications costs per retrieved oocyte | Ten to fifteen days after starting ovarian stimulation]
  Total cost of medications used in all cycles/number of retrieved oocytes

SECONDARY OUTCOMES:
Clinical pregnancy rate | 5 weeks after embryo transfer]
  Presence of intrauterine gestational sac detected by transvaginal ultrasound
Ongoing Pregnancy Rate | 18 weeks after embryo transfer]
  Pregnancies continued beyond 20 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Aboul Foutouh, Prof., Study Chair — Cairo University
Locations (1):
- Bedaya Hospital, Giza, Egypt

REFERENCES:
- [Background] Ubaldi FM, Capalbo A, Vaiarelli A, Cimadomo D, Colamaria S, Alviggi C, Trabucco E, Venturella R, Vajta G, Rienzi L. Follicular versus luteal phase ovarian stimulation during the same menstrual cycle (DuoStim) in a reduced ovarian reserve population results in a similar euploid blastocyst formation rate: new insight in ovarian reserve exploitation. Fertil Steril. 2016 Jun;105(6):1488-1495.e1. doi: 10.1016/j.fertnstert.2016.03.002. Epub 2016 Mar 25. PMID 27020168